CLINICAL TRIAL: NCT05938569
Title: Computer-Assisted Hair Restoration Study Using ARTAS System
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-017
Record Dates: First submitted 2023-06-27; First posted 2023-07-10 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- All subjects (Experimental): The Study Treatment will involve follicular hair unit harvest, recipient site making, and implantation.
  Interventions: Device: Hair restoration

INTERVENTIONS:
Device: Hair restoration — The Study Treatment will involve follicular hair unit harvest, recipient site making, and implantation.

SUMMARY:
Prospective, multi-center, up to 4 investigational centers evaluating the performance of the ARTAS System in Hair Restoration Procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male with clinical diagnosis of androgenetic alopecia with Norwood-Hamilton grade of III-VI
* Subject is 20 to 70 years old
* Subject agrees to cut hair short (< 1 mm) on the scalp in the designated study areas for harvesting and implantation
* Subject is able to understand and provide written consent
* Subject consents to post-operative follow-up per protocol

Exclusion Criteria:

* Subject has prior history of scalp reduction surgery(s) in the past six months
* Subject has bleeding diathesis
* Subject has active use of anti-coagulation medication
* Subject has any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study

Ages: 20 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11-03; Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in Hair Density from pre to 12 months post-treatment in robotic vs manual implantation | 1 year post-treatment

SECONDARY OUTCOMES:
Percentage of follicles successfully harvested by Robot | 1 year post-treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Berman Skin Institute, Los Altos, California
  - Le's Aesthetics, San Jose, California

IPD SHARING:
Plan to Share IPD: No